CLINICAL TRIAL: NCT01759420
Title: Ondansetron and the QT Interval In Adult Emergency Department Patients
Status: Completed | Type: Observational
Sponsor: C.R.Darnall Army Medical Center (U.S. Federal Agency)
Collaborators: Madigan Army Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Peter Moffett MD, Director of Research, Department of Emergency Medicine, C.R.Darnall Army Medical Center
Other Study IDs: 375393
Record Dates: First submitted 2012-12-29; First posted 2013-01-03 (Estimated); Results first posted 2014-06-26 (Estimated); Last update posted 2014-06-26 (Estimated); Status verified 2014-06

CONDITIONS: Ondansetron
Keywords: Ondansetron; QT interval; QTc; QT prolongation; Drug induced QT prolongation
MeSH Terms: conditions — Long QT Syndrome | interventions — Ondansetron

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- IV Ondansetron: Adult emergency department patients receiving 4mg of IV ondansetron as part of their treatment plan.
  Interventions: Drug: Ondansetron

INTERVENTIONS:
Drug: Ondansetron — 4mg of intravenous ondansetron
  Other Names: Zofran

SUMMARY:
The purpose of this study is to assess the use of the medication ondansetron (zofran) in the emergency department. There are studies of the ability of ondansetron to cause a prolongation in the QT interval (a certain measurement on an EKG) in anesthesia and cancer patients, but not on emergency department patients. This is an observational study where patients that are going to receive the anti-nausea medicine ondansetron in the emergency department will have an EKG performed every 2 minutes for 20 minutes to determine if the QT interval prolongs and returns to normal in that time period. Any serious outcomes will be reported. There is expected to be no adverse outcomes from this routinely used medication.

DETAILED DESCRIPTION:
Intravenous ondansetron is routinely used in adult emergency department patients experiencing nausea or vomiting. The FDA has changed the drug label to warn of prolongation of the QT interval and required the manufacturer to perform additional studies. There are rare case reports of cardiac electrical toxicity to include QT prolongation, atrial fibrillation, severe bradycardia, ventricular tachycardia, supraventricular tachycardia, and the potential for Torsades de Pointes. All of the reported literature on ondansetron comes from post-operative patients, patients receiving chemotherapy, and healthy volunteers, but has never been assessed in the emergency department population. Adult emergency department patients that do not meet the exclusion criteria will be enrolled prior to receiving intravenous ondansetron. Administration of ondansetron will be at the discretion of the attending physician. A twelve-lead electrocardiogram (EKG) or 12-lead rhythm strip will be generated prior to drug administration, and every 2 minutes following drug administration for 20 minutes after administration. During the entire 20 minutes the patient will be on a cardiac monitor and if any of the defined adverse cardiac electrical events occur (non-sinus rhythm, severe bradycardia, sudden cardiac death) the patient will be treated using standard Advanced Cardiac Life Support methods and admitted for continued monitoring. The mean maximal QTc prolongation (as measured by the Bazett formula), as well as the rate of adverse cardiac events with 95% confidence intervals will be reported.

The global objective of this study is to determine if routine use of intravenous ondansetron in the emergency department is associated with cardiac risks. The primary objective is to determine the mean maximal prolongation in QTc interval from baseline as measured by the Bazett formula. The secondary objective is to determine the number of severe adverse cardiac electrical events (non-sinus rhythm, severe bradycardia, sudden cardiac death) associated with routine use of intravenous ondansetron in the adult emergency department patient.

ELIGIBILITY:
Inclusion Criteria:

* Age >18
* Patient to receive 4mg of intravenous ondansetron

Exclusion Criteria:

* Age <18
* known long QT syndrome
* received oral or intravenous ondansetron within 4 hours of enrollment
* co-administration of any known QT prolonging agents
* QTc on baseline of >450 ms for males and >470ms for females
* allergy or known hypersensitivity to ondansetron
* altered mental status
* non-sinus rhythm on baseline EKG
* hypokalemia (as defined by the lower limit of normal for the reference laboratory)
* hypomagnesemia (as defined by the lower limit of normal for the reference laboratory)
* any presentation for chest pain with signs of ischemia on baseline EKG
* QRS duration > 120 msec
* bundle branch block (right or left)
* ventricular pre-excitation or signs of left ventricular hypertrophy with repolarization abnormalities

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The target population is adult (>18 years old) emergency department patients who have been deemed appropriate to receive intravenous ondansetron.
Sampling Method: Non-Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2012-12; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter M Moffett, MD, Principal Investigator — Carl R Darnall Army Medical Center Department of Emergency Medicine
Locations (2):
- United States (2):
  - Carl R Darnall Army Medical Center, Fort Hood, Texas
  - Madigan Army Medical Center, Tacoma, Washington

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | IV Ondansetron
Started | 28
Completed | 22
Not Completed | 6
Not completed — Screen failure | 5
Not completed — Inaccurate EKG machine readings | 1

BASELINE CHARACTERISTICS:
Arm/Group | IV Ondansetron
Number analyzed (Participants) | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 22
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 9

OUTCOME MEASURES:

1. Primary Outcome: Change in QTc Interval With Ondansetron Administration
Description: The primary objective is to determine the mean maximal prolongation in QTc interval from baseline as measured by the Bazett formula. A baseline EKG will be obtained and then after drug administration an EKG will be performed every 2 minutes until 20 minutes has passed. The mean maximal QTc change will be calculated.
Time Frame: Baseline to 20 minutes
Measure: Mean (95% Confidence Interval); unit: mS
Arm/Group | IV Ondansetron
Number analyzed (Participants) | 22
mS | 19.7 [14 to 25.5]

2. Secondary Outcome: Number of Adverse Events
Description: The secondary objective is to determine the number of severe adverse cardiac electrical events (non-sinus rhythm, severe bradycardia, sudden cardiac death) associated with routine use of intravenous ondansetron in the adult emergency department patient. All of these outcomes will be recorded for each patient during the emergency department stay which could range from 20 minutes to several hours.
Time Frame: 20 minutes to 8 hours
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | IV Ondansetron
Number analyzed (Participants) | 23
percentage of patients | 0 [0 to 12.5]

ADVERSE EVENTS:
Arm/Group | IV Ondansetron
Serious Adverse Events (participants affected / at risk) | 0/23
Other Adverse Events (participants affected / at risk) | 0/23

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes